CLINICAL TRIAL: NCT02047136
Title: Can Low Histamine Diet Reduce Symptoms of Patients With Idiopathic Urticaria?
Brief Title: Dietary Treatment for Chronic Urticaria
Acronym: DTCU
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to recruit subjects, patients want active treatment instead of placebo.
Sponsor: Hong Kong Sanatorium & Hospital (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ALC-001
Record Dates: First submitted 2014-01-24; First posted 2014-01-28 (Estimated); Last update posted 2018-08-02 (Actual); Status verified 2018-07

CONDITIONS: Diet Modification; Chronic Urticaria
MeSH Terms: conditions — Chronic Urticaria

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment group (on low histamine diet) (Experimental): 78 subjects who come to Allergy Centre for treatment of idiopathic urticaria, with or without angioedema and pruritus (U/A/P), will be randomized into two parallel groups; treatment group (TG) will be asked to follow a histamine-restricted diet for 4 weeks and the control group (CG) will be asked to follow a well-balanced diet instructed by a dietitian for 4 weeks. A well-balanced diet for the CG subject is tailor-made by the dietitian according to subject's usual intake to ensure that the subject's energy requirement is met and all food groups are consumed.
  Interventions: Other: Treatment group (on low histamine diet)
- Well-balanced diet (Active Comparator): Diet tailor-made by the dietitian according to subject's usual intake to ensure that the subject's energy requirement is met and all food groups are consumed.
  Interventions: Other: Well-balanced diet

INTERVENTIONS:
Other: Treatment group (on low histamine diet) — 78 subjects who come to Allergy Centre for treatment of idiopathic urticaria, with or without angioedema and pruritus (U/A/P), will be randomized into two parallel groups; treatment group (TG) will be asked to follow a histamine-restricted diet for 4 weeks and the control group (CG) will be asked to follow a well-balanced diet instructed by a dietitian for 4 weeks. A well-balanced diet for the CG subject is tailor-made by the dietitian according to subject's usual intake to ensure that the subject's energy requirement is met and all food groups are consumed.
  Arms: Treatment group (on low histamine diet)
Other: Well-balanced diet — Diet tailor-made by the dietitian according to subject's usual intake to ensure that the subject's energy requirement is met and all food groups are consumed.
  Arms: Well-balanced diet

SUMMARY:
Histamine is a biologically active component that can be found in many foods and beverages. Intake of excessive histamine from foods or beverages, can trigger symptoms including urticaria. A low histamine diet has been recommended as one of the possible treatments for patients with chronic urticaria. There are very few studies to confirm the effectiveness of such diets and, to the investigators' knowledge, none from Asia where high histamine containing meals are often eaten (personal observations). The objective of the present study is to investigate the therapeutic effect of low histamine diet in relieving symptoms in patients with chronic urticaria with or without angioedema, and / or pruritus (U/A/P). The investigators hypothesize that following a low histamine diet for 4 weeks, the symptoms of patients with chronic U/A/P should improve.

DETAILED DESCRIPTION:
A double blinded parallel randomized control study over 4 weeks will be conducted to assess the effectiveness of a histamine-restricted diet. Neither the subjects nor the medical investigator will know which diet is being prescribed.

The study will only be conducted after ethical approval has been granted and with informed consent. If it is a child, informed consent will be obtained from a parent. Subject has to pay his/her consultation fee for doctor's and dietitian's consultation and skin prick and/or blood tests at the first visit as normal but there will be no charge for subsequent visits in relation to the trial.

A period of 4 weeks on the low histamine diet has previously been shown to be sufficient to determine whether dietary manipulation will help in the management of the urticaria symptoms.

Selection Criteria and sample size calculation 78 subjects who come to Allergy Centre for treatment of idiopathic urticaria, with or without angioedema and pruritus (U/A/P), will be randomized into two parallel groups; treatment group (TG) will be asked to follow a histamine-restricted diet for 4 weeks and the control group (CG) will be asked to follow a well-balanced diet instructed by a dietitian for 4 weeks. A well-balanced diet for the CG subject is tailor-made by the dietitian according to subject's usual intake to ensure that the subject's energy requirement is met and all food groups are consumed. Subjects in both groups are also instructed to have adequate water intake during the study period. Both groups are asked to record food diary and symptoms during the study period. Consent form will state that it is a study to compare the efficacy of both diets. After the study period, subjects in the CG will be able to follow a low histamine diet if this is proven to be beneficial, so everyone will have the potential to benefit from the low histamine diet and vice versa for the TG subjects.

Low Histamine Diet Histamine is present in almost all foods in small quantities. Its presence increases with maturation of the food. High quantities of histamine are found mainly in products of microbial fermentation, such as aged cheese, sauerkraut, wine, and processed meat. Some oriental foods with high histamine content are also included.The current Low Histamine Diet sheet of Hong Kong Sanatorium & Hospital will be used (Appendix I).

Evaluation of Symptoms When a subject comes for the first consultation (randomization week), he/she will be given a 4-point scale questionnaire (see Appendix II) to evaluate his/her own symptoms (pruritus severity and number of wheals). This will be completed once every evening for a week prior to the 4-week treatment period. The pruritus severity score and the number of wheals during this run in week will be averaged and used as the mean baseline score. The summation of mean pruritus score (MPS) and the mean number of wheals (MNW) will be the mean total symptoms score (MTSS) for the baseline period. Medical investigator will also evaluate the subject's global symptoms severity (GSS) at the first consultation (randomization week) and second consultation (at the end of week 4).

MPS and GSS is scored as 0 = none; 1 = mild (present but not disturbing); 2 = moderate (disturbing but not hampering day time activities and/or sleep); and 3 = severe/intense (disturbing and hampering day time activities and/or sleep). Number of wheals are scored as 0 = none; 1 = mild (less than 20 wheals per 24 hours); 2 = moderate (21-50 wheals); and 3 = severe (more than 50 wheals).

After the first consultation with the medical investigator, a skin prick test and/or blood tests for specific immunoglobulin E (IgE) to eight major food allergens will be tested, namely cow's milk, egg, peanut, treenuts, wheat, soya, seafood, shellfish. Subject will consult a dietitian for either a well-balanced diet (CG) or low histamine diet (TG) and he/she is asked only to start the diet one week after the first consultation. The subject will be asked to fax or email his/her completed questionnaire and food diary for checking before he/she starts the diet. Dietitian will ensure that the questionnaire and the food diary are completed correctly by the subject. Dietitian will then phone the subject not only to remind him/her to start on the diet but also to make sure that the subject corrects any errors in completing the questionnaire and food diary. If the diary during the run in period is done very poorly it may have to be repeated before the formal diet begins. Dietitian will conduct subsequent weekly phone follow up with each subject. Each subject will be reminded to complete their questionnaires and food diaries every evening.

For each symptom the scores for each week will be averaged. The sum of MPS and MNW is the mean total symptoms score (MTSS) and this will also be averaged for each week period.

Evaluation of compliance of low histamine diet

Each subject will complete a food diary, in addition to the symptom score chart, where he/she will record his/her dietary intake for each snack and meal during the 4-week study period. The food diary will be evaluated by the Allergy Centre dietitians for adherence to the diet. Diet compliance score (DCS) is scored as 0 = not comply at all; 1 = poor diet compliance (intake of 2 or more high histamine foods daily); 2 = good compliance (intake of 1 or less high histamine food daily); 3 = excellent diet compliance (intake of 3 or less high histamine food per week).

Randomization and blinding After provision of informed consent, subjects will be allocated by a table of random numbers to either the TG or CG. The number sequence will be generated by the computer list prepared by dietitians. Neither the subjects nor the medical investigator will know which diet is being prescribed to which subject.

Power calculations and statistical analysis

Sample size was determined based on a previous drug study13 as there is insufficient data on low histamine diets. To detect a clinically significant mean difference of at least 1 point between the active and control groups on the 4 point scale with 80% power at p< 0.05 requires 35 subjects in each trial arm. Allowing for a 10% drop out rate, the total sample should be 78 individuals.

Statistical analyses will be performed by hospital statisticians using SPSS version 18.0.0 (2009). The primary outcomes will be the change in Mean Total Symptoms Score (MTSS) from baseline between groups. Secondary outcome measures will include assessment of (1) the change in MPS between groups; (2) the change in MNW between groups. (3) the change in GSS by medical investigator between groups; (4) the comparison of area under the curve (AUC for the trend) for MTSS, MPS, MNW, GSS and DCS between the groups during the 4-week period; and (5) the comparison of total dose of anti-histamine used by each group compared to baseline within the study period. All data will be analyzed using paired student's t-test.

ELIGIBILITY:
Inclusion Criteria:

* Urticaria +/- angioedema present for a minimum of 6 weeks;
* Agree to be on anti-histamine prn;
* Age older than 8 years old, with no upper age limit;
* Causes such as parasite infestation, microbial and viral infections, autoimmune disease, or other pathology that could account for the U/A/P should be excluded;
* Skin prick test and/or radioallergosorbent (RAST) test are negative for all food allergens tested, or patient had achieved no symptomatic improvement after strict avoidance of all skin test-positive foods;

Exclusion Criteria:

* Pregnant or breast feeding women;
* Patients who is taking central nervous system (CNS) acting agents (including tranquilizers, antidepressants, sedatives, hypnotics or antiepileptics) at any time;

Min Age: 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
The change in Mean Total Symptoms Score (MTSS) from baseline between groups | 4 weeks
  When a subject comes for the first consultation (randomization week), he/she will be given a 4-point scale questionnaire (see Appendix II) to evaluate his/her own symptoms (pruritus severity and number of wheals). This will be completed once every evening for a week prior to the 4-week treatment period. The pruritus severity score and the number of wheals during this run in week will be averaged and used as the mean baseline score. The summation of mean pruritus score (MPS) and the mean number of wheals (MNW) will be the mean total symptoms score (MTSS) for the baseline period. Then comparison between the change in Mean Total Symptoms Score (MTSS) from baseline between treatment group and control group.

SECONDARY OUTCOMES:
the change in mean pruritus score (MPS) between treatment group and control group | 4 week
  When a subject comes for the first consultation (randomization week), he/she will be given a 4-point scale questionnaire (see Appendix II) to evaluate his/her own symptoms (pruritus severity and number of wheals). This will be completed once every evening for a week prior to the 4-week treatment period. The pruritus severity score and the number of wheals during this run in week will be averaged and used as the mean baseline score. The summation of mean pruritus score (MPS) and the mean number of wheals (MNW) will be the mean total symptoms score (MTSS) for the baseline period.
the change in mean number of wheals (MNW) between groups | 4 week
  When a subject comes for the first consultation (randomization week), he/she will be given a 4-point scale questionnaire to evaluate his/her own symptoms (pruritus severity and number of wheals). This will be completed once every evening for a week prior to the 4-week treatment period. The pruritus severity score and the number of wheals during this run in week will be averaged and used as the mean baseline score. The summation of mean pruritus score (MPS) and the mean number of wheals (MNW) will be the mean total symptoms score (MTSS) for the baseline period.
the change in global symptoms severity (GSS) by medical investigator between groups | 5 weeks
  Medical investigator will also evaluate the subject's global symptoms severity (GSS) at the first consultation (randomization week) and second consultation (at the end of week 4).
the comparison of area under the curve (AUC for the trend) for MTSS, MPS, MNW, GSS and DCS between the groups during the 4-week period | 4 week
  When a subject comes for the first consultation (randomization week), he/she will be given a 4-point scale questionnaire to evaluate his/her own symptoms (pruritus severity and number of wheals). This will be completed once every evening for a week prior to the 4-week treatment period. The pruritus severity score and the number of wheals during this run in week will be averaged and used as the mean baseline score. The summation of mean pruritus score (MPS) and the mean number of wheals (MNW) will be the mean total symptoms score (MTSS) for the baseline period. Medical investigator will also evaluate the subject's global symptoms severity (GSS) at the first consultation (randomization week) and second consultation (at the end of week 4).
  MPS and GSS is scored as 0 = none; 1 = mild (present but not disturbing); 2 = moderate (disturbing but not hampering day time activities and/or sleep); and 3 = severe/intense (disturbing and hampering day time activities and/or sleep).

CONTACTS AND LOCATIONS:
Overall Officials: Wai Yan Vivian Lau, Master, Principal Investigator — Hong Kong Sanatorium & Hospital
Locations (1):
- Hong Kong Sanatorium & Hospital, Hong Kong, China

REFERENCES:
- [Result] Maintz L, Novak N. Histamine and histamine intolerance. Am J Clin Nutr. 2007 May;85(5):1185-96. doi: 10.1093/ajcn/85.5.1185. PMID 17490952
- [Result] Janice M. Vickerstaff Joneja, Cabrini Carmona-Silva. Outcome of a Histamine-restricted Diet Based on Chart Audit. Journal of Nutritional and Environmental Medicine 11(4): 249-262, 2001.